CLINICAL TRIAL: NCT02549170
Title: A Phase III Study to Evaluate the Efficacy, Safety, and Tolerability of Immune Globulin Infusion 10% (Human) With Recombinant Human Hyaluronidase (HYQVIA/HyQvia) and Immune Globulin Infusion (Human), 10% (GAMMAGARD LIQUID/KIOVIG) for the Treatment of Chronic Inflammatory Demyelinating Polyradiculoneuropathy (CIDP)
Brief Title: A Study of HyQvia and Gammagard Liquid (Kiovig) in Adults With Chronic Inflammatory Demyelinating Polyradiculoneuropathy (CIDP)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Baxalta now part of Shire (Industry)
Collaborators: Takeda Development Center Americas, Inc. (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 161403; 2014-005496-87 (EudraCT Number)
Record Dates: First submitted 2015-09-11; First posted 2015-09-15 (Estimated); Results first posted 2023-05-24 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Chronic Inflammatory Demyelinating Polyradiculoneuropathy
Keywords: Autoimmune Diseases; Polyneuropathies; Nervous System Diseases; Peripheral Nervous System Diseases; Polyradiculoneuropathy; Autoimmune Diseases of the Nervous System; Immunoglobulins; Immune System Diseases; Demyelinating Diseases; Polyradiculoneuropathy, Chronic Inflammatory Demyelinating; Neuromuscular Diseases
MeSH Terms: conditions — Polyradiculoneuropathy, Chronic Inflammatory Demyelinating; Autoimmune Diseases; Polyneuropathies; Nervous System Diseases; Peripheral Nervous System Diseases; Polyradiculoneuropathy; Autoimmune Diseases of the Nervous System; Immune System Diseases; Demyelinating Diseases; Neuromuscular Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Epoch 1: HYQVIA/HyQvia (Experimental): Participants received HYQVIA/HyQvia (rHuPH20) 80 U/g IG, following by SC injection of immunoglobulin (IGI) 10% at the same monthly equivalent IG dose as the individual participant's pre-randomized IG dose when administered every 2, 3, or 4 weeks for 30.28 weeks or until relapse.
  Interventions: Biological: HYQVIA
- Epoch 1: Placebo with rHuPH20 (Placebo Comparator): Participants received rHuPH20 80 U/I0 mL placebo solution, followed by SC placebo infusion at matching infusion volume as the participant's pre-randomization monthly equivalent IG dose when administered every 2, 3, or 4 weeks for 31.54 weeks or until relapse.
  Interventions: Biological: 0.25% albumin placebo solution with rHuPH20
- Epoch 2: E1: Placebo Relapse - E2: GGL/KIOVIG (Experimental): Participants who were enrolled to receive placebo with rHuPH20 and achieved chronic inflammatory demyelinating polyradiculoneuropathy (CIDP) relapse during Epoch 1 received the induction dose of GGL/KIOVIG 2 g/kg bi-weekly (BW), followed by IV infusion at the same monthly equivalent dose as the participant's pre-randomization IGIV dosing regimen when administered every 3 weeks for 25.63 weeks or until relapse.
  Interventions: Biological: IGIV GAMMAGARD LIQUID/KIOVIG
- Epoch 2: E1: HYQVIA Relapse - E2: GGL/KIOVIG (Experimental): Participants who were enrolled to receive HYQVIA/HyQvia (rHuPH20) and achieved CIDP relapse during Epoch 1 received the induction dose of GGL/KIOVIG 2 g/kg BW, followed by IV infusion at the same monthly equivalent dose as the participant's pre-randomization IGIV dosing regimen when administered every 3 weeks for 28.67 weeks or until relapse.
  Interventions: Biological: IGIV GAMMAGARD LIQUID/KIOVIG
- Epoch 2: E1: Placebo Relapse - E2: GAMMUNEX-C (Experimental): Participants who were enrolled to receive placebo with rHuPH20 and achieved CIDP relapse during Epoch 1 received the induction dose of GAMMUNEX-C 2 g/kg BW, followed by IV infusion at the same monthly equivalent dose as the participant's pre-randomization IGIV dosing regimen when administered every 3 weeks for 24.33 weeks or until relapse.
  Interventions: Biological: IGIV GAMUNEX®-C

INTERVENTIONS:
Biological: HYQVIA — Participants will receive HYQVIA/HyQvia SC which contains both Immune Globulin Infusion 10% (Human) (IGI, 10%) and recombinant human hyaluronidase (rHuPH20).
  Other Names: 10%) with recombinant human hyaluronidase (rHuPH20); Immune Globulin Infusion 10% (Human) (IGI; IGI; 10% with rHuPH20
  Arms: Epoch 1: HYQVIA/HyQvia
Biological: 0.25% albumin placebo solution with rHuPH20 — Participants will receive placebo solution (0.25% human albumin in Lactated Ringer's solution) and rHuPH20.
  Arms: Epoch 1: Placebo with rHuPH20
Biological: IGIV GAMMAGARD LIQUID/KIOVIG — Participants will receive GAMMAGARD LIQUID/KIOVIG
  Other Names: Immune Globulin Infusion (Human); Intravenous immunoglobulin G; 10% (GAMMAGARD LIQUID/KIOVIG); GAMMAGARD LIQUID
  Arms: Epoch 2: E1: HYQVIA Relapse - E2: GGL/KIOVIG; Epoch 2: E1: Placebo Relapse - E2: GGL/KIOVIG
Biological: IGIV GAMUNEX®-C — Participants will receive GAMUNEX®-C
  Other Names: Immune Globulin Infusion (Human); Intravenous immunoglobulin G; Approved IGIV product for US sites
  Arms: Epoch 2: E1: Placebo Relapse - E2: GAMMUNEX-C

SUMMARY:
The aim of this study is to learn more about the following treatment options in adults with CIDP:

* Subcutaneous self-infusion with HyQvia.
* Intravenous infusion with Gammagard/Kiovig. Gammagard and Kiovig are the brand names for the same immunoglobulin compound.

The study is in two parts. In Part 1, participants receive either HyQvia or a placebo subcutaneously. In Part 2 (only for participants who have a CIPD relapse during Part 1), participants will receive Gammagard Liquid/Kiovig intravenously. US participants will receive Gamunex-C.

The first SC infusion will be given in the study clinic. The remaining SC infusions may be given in the study clinic or the participant's home. This will be decided by the study doctor and whether the participant or their caregiver can do the self-infusion.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females of age greater than or equal to (>=)18 years old at the time of screening.
2. Participant has a documented diagnosis of definite or probable Chronic inflammatory demyelinating polyradiculoneuropathy (CIDP) (focal atypical CIDP and pure sensory atypical CIDP will be excluded), as confirmed by a neurologist specializing/experienced in neuromuscular diseases to be consistent with the European Federation of Neurological Societies/Peripheral Nerve Society (EFNS/PNS) 2010 criteria (European Federation of Neurological Societies, 2010). Fulfillment of electrodiagnostic criteria must be confirmed by an independent qualified/experienced central reader.
3. Participant has responded to IgG treatment in the past (partial or complete resolution of neurological symptoms and deficits), and must currently be on stable doses of IGIV treatment within the dose range equivalent to a cumulative monthly dose of 0.4 to 2.4 gram per kilogram (g/kg) BW (inclusive) administered intravenously for at least 12 weeks prior to screening. The dosing interval of IGIV treatment must be between 2 and 6 weeks (inclusive). Variations in the dosing interval of up to ± 7 days or monthly dose amount of up to ± 20% between participant's pre-study Immunoglobulin G (IgG) infusions are within acceptable limits.
4. INCAT disability score between 0 and 7 (inclusive). Participants with INCAT scores of 0, 1 (whether from upper or lower extremities), or 2 (if at least 1 point is from an upper extremity) at screening and/or baseline will be required to have a history of significant disability as defined by an INCAT disability score of 2 (must be exclusively from the lower extremities) or greater documented in the medical record. Participants will be eligible if one of the below eligibility criteria are met:

   Screening and Baseline INCAT disability score of between 3 and 7 inclusive.
   1. Screening and/or Baseline INCAT disability score of 2 (both points are from lower extremities).
   2. Screening and/or Baseline INCAT disability score of 2 (both points are not from lower extremities) AND has at least a score of 2 or greater documented in the medical record prior to screening. If a score was greater than 2 documented in the medical record prior to screening at least 2 points must be from lower extremities.
   3. Screening and/or Baseline INCAT disability score of 0 or 1 AND has at least a score of 2 or greater (both from lower extremities) documented in the medical record prior to screening, at least 2 points must be from lower extremities.
5. If female of childbearing potential, the participant must have a negative pregnancy test at screening and agree to employ a highly effective contraceptive measure throughout the course of the study and for at least 30 days after the last administration of investigational product (IP).
6. Participant is willing and able to sign an Informed Consent Form (ICF).
7. Participant is willing and able to comply with the requirements of the protocol.

Exclusion Criteria:

1. Participants with Focal atypical CIDP or pure sensory atypical CIDP.
2. Any neuropathy of other causes, including:

   1. Hereditary demyelinating neuropathies, such as hereditary sensory and motor neuropathy (HSMN) (Charcot-Marie-Tooth [CMT] disease), and hereditary sensory and autonomic neuropathies (HSANs).
   2. Neuropathies secondary to infections, disorders, or systemic diseases such as Borrelia burgdorferi infection (Lyme disease), diphtheria, systemic lupus erythematosus, POEMS (polyneuropathy, organomegaly, endocrinopathy, M-protein, and skin changes) syndrome, osteosclerotic myeloma, diabetic and non-diabetic lumbosacral radiculoplexus neuropathy, lymphoma, and amyloidosis.
   3. Multifocal acquired demyelinating sensory and motor neuropathy (MADSAM).
   4. Multifocal motor neuropathy (MMN).
   5. Drug-, biologic-, chemotherapy-, or toxin-induced peripheral neuropathy.
3. Immunoglobulin M (IgM) paraproteinemia, including IgM monoclonal gammopathy with high titer antibodies to myelin-associated glycoprotein.
4. Prominent sphincter disturbance.
5. Central demyelinating disorders (eg, multiple sclerosis).
6. Any chronic or debilitating disease, or central nervous disorder that causes neurological symptoms or may interfere with assessment of CIDP or outcome measures (eg, arthritis, stroke, Parkinson's disease, and diabetic peripheral neuropathy) (Participants with clinically diagnosed diabetes mellitus who do not have diabetic peripheral neuropathy, who have adequate glycemic control with Hemoglobin A1C; also known as glycosylated or glycated hemoglobin (HbA1C) of less than (<) 7.5% at screening, and who agree to maintain adequate glycemic control during the study are allowed).
7. Congestive heart failure (New York Heart Association [NYHA] Class III/IV), unstable angina, unstable cardiac arrhythmias, or uncontrolled hypertension (ie, diastolic blood pressure greater than (>) 100 millimeter of mercury (mmHg) and/or systolic blood pressure >160 mmHg).
8. History of deep vein thrombosis or thromboembolic events (eg, cerebrovascular accident, pulmonary embolism) in the past 12 months.
9. Condition(s) which could alter protein catabolism and/or IgG utilization (eg, protein-losing enteropathies, nephrotic syndrome).
10. Known history of chronic kidney disease, or glomerular filtration rate (GFR) of <60 milliliter per minute per 1.73 square meter (mL/min/1.73m^2) estimated based on CKD-EPI equation (Levey et al., 2009) at the time of screening.
11. Participant with active malignancy requiring chemotherapy and/or radiotherapy, or history of malignancy with less than 2 years of complete remission prior to screening. Exceptions are: adequately treated basal cell or squamous cell carcinoma of the skin, carcinoma in situ of the cervix, and stable prostate cancer not requiring treatment.
12. Clinically significant anemia or hemoglobin (Hgb) level of less than (<) 10.0 grams per deciliter (g/dL) at screening.
13. Hypersensitivity or adverse reactions (AR's) (eg, urticaria, breathing difficulty, severe hypotension, or anaphylaxis) to human blood products such as human IgG, albumin, or other blood components.
14. Known allergy to hyaluronidase of human (including recombinant human hyaluronidase) or animal origin (such as bee or wasp venom).
15. Known history of or immunoglobulin A (IgA) deficiency (<8 milligram per deciliter [mg/dL]) at screening.
16. Abnormal laboratory values at screening:

    1. Serum aspartate aminotransferase (AST) and alanine aminotransferase (ALT) > 2.5* upper limit of normal (ULN)
    2. Platelet count <100,000 cells per microliter (cells/mcL).
    3. Absolute neutrophil count (ANC) <1000 cells/mcL.
17. Ongoing/active infection with hepatitis A virus (HAV), hepatitis B virus (HBV), hepatitis C virus (HCV), or human immunodeficiency virus (HIV) Type 1/2 infection.
18. The participant has received or is currently receiving treatment with immunomodulatory/ immunosuppressive agents within 6 months prior to screening.
19. Participant has received or is currently receiving treatment with corticosteroids dose within 8 weeks prior to screening, regardless of indication.
20. Participant has undergone plasma exchange (PE) within 3 months prior to screening.
21. The participant has any disorder or condition that in the investigator's judgment may impede the participant's participation in the study, pose increased risk to the participant, or confound the results of the study.
22. The participant is nursing or intends to begin nursing during the course of the study.
23. Participant has participated in another clinical study involving an IP or investigational device within 30 days prior to enrollment, or is scheduled to participate in another clinical study (with the exception of the HYQVIA/HyQvia extension study in CIDP) involving an IP or investigational device during the course of this study.
24. The participant is a family member or employee of the investigator.
25. Participants with acquired or inherited thrombophilic disorders. These will include the specific types of acquired or inherited thrombophilic disorders that could put participants at risk of develop thrombotic events. Examples include:

    a. Hereditary Thrombophilias i. Factor V Leiden mutation. ii. Prothrombin 20210A mutation. iii. Protein C deficiency. iv. Protein S deficiency. v. Antithrombin deficiency. b. Acquired thrombophilias i. Antiphospholipid antibody syndrome. ii. Activated protein C Resistance acquired. iii. Homocystinemia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2015-12-15 (Actual); Primary Completion 2022-02-23 (Actual); Study Completion 2022-02-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Shire
Locations (83):
- United States (19):
  - Barrow Neurological Institute, Phoenix, Arizona
  - Arizona Neuromuscular Research Center, Phoenix, Arizona
  - HonorHealth Neurology, Scottsdale, Arizona
  - University of California-Irvine, Orange, California
  - Forbes Norris Mda/als Ctr, San Francisco, California
  - Regents of the University of colorado, Aurora, Colorado
  - Immunoe Research Centers, Centennial, Colorado
  - University of South Florida, Tampa, Florida
  - University of Kansas Medical Center Research Institute, Inc., Kansas City, Kansas
  - William Beaumont Hospital, Royal Oak, Michigan
  - Neurology Center of Las Vegas, Las Vegas, Nevada
  - Rutgers New Jersey Medical School, Newark, New Jersey
  - Hospital for Special Surgery, New York, New York
  - Wake Forest University, Winston-Salem, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Austin Neuromuscular Center, Austin, Texas
  - The Methodist Hospital Research Institute, Houston, Texas
  - University Texas Physicians CAR, Houston, Texas
- Argentina (4):
  - Hospital Italiano, Ciudad Autonoma Buenos Aires, Buenos Aires
  - Hospital Britanico de Buenos Aires, Ciudad Autonoma Buenos Aires
  - Complejo Medico de la Policia Federal Argentina Churruca Visca, Ciudad Autonoma Buenos Aires
  - Instituto de Investigaciones Neurologicas Raul Carrea, FLENI, Ciudad Autonoma Buenos Aires
- Brazil (5):
  - Instituto de Neurologia de Curitiba - Hospital Ecoville, Curitiba, Paraná
  - HUAP - UFF - Hospital Universitario Antonio Pedro - Universidade Federal Fluminense, Niterói, Rio Do Janeiro
  - Hospital das Clínicas da Faculdade de Medicina da UNICAMP, Campinas, São Paulo
  - Hospital das Clínicas FMRP-USP, Ribeirão Preto, São Paulo
  - Hospital Sao Paulo, São Paulo, São Paulo
- Canada (3):
  - University of Alberta Hospital, Edmonton, Alberta
  - LHSC - University Hospital, London, Ontario
  - Toronto General Hospital, Toronto, Ontario
- Institucion Prestadora de Servicios de Salud de la Universidad de Antioquia "IPS UNIVERSITARIA", Medellín, Colombia
- Croatia (3):
  - Clinical Hospital Centre Rijeka, Rijeka
  - Clinical Hospital Centar Zagreb, Zagreb
  - University Hospital Centre "Sestre Milosrdnice", Zagreb
- Czechia (3):
  - Fakultni nemocnice Brno, Brno
  - Fakultni nemocnice Ostrava, Ostrava - Poruba
  - Fakultni nemocnice v Motole, Prague
- Århus Universitetshospital, Aarhus, Denmark
- France (4):
  - CHU de Nice Hôpital Pasteur 2, Nice, Alpes Maritimes
  - Hôpital de la Timone, Marseille, Bouches-du-Rhône
  - Groupe Hospitalier Pellegrin - Hôpital Pellegrin, Bordeaux, Gironde
  - Hopital Neurologique Pierre Wertheimer, Bron, Rhone
- Germany (3):
  - Universitaetsmedizin Goettingen, Göttingen, Lower Saxony
  - Universitaetsklinikum Essen, Essen, North Rhine-Westphalia
  - Universitaetsklinikum Leipzig AoeR, Leipzig, Saxony
- University Hospital of Patra, Pátrai, Greece
- Chaim Sheba Medical Center, Ramat Gan, Israel
- Italy (11):
  - IRCCS Ospedale Casa Sollievo della Sofferenza, San Giovanni Rotondo, Foggia
  - Istituto Clinico Humanitas, Rozzano, Milano
  - Azienda Ospedaliera Universitaria Policlinico Tor Vergata, Rome, Roma
  - Azienda Ospedaliero Universitaria San Martino, Genova
  - Azienda Ospedaliera Universitaria Policlinico G. Martino, Messina
  - Casa di Cura del Policlinico, Milan
  - Fondazione Istituto Neurologico Casimiro Mondino, Pavia
  - Azienda Ospedaliero Universitaria Pisana, Pisa
  - Azienda Ospedaliera Universitaria Policlinico Umberto I - Università di Roma La Sapienza, Roma
  - Azienda Ospedaliera Città della Salute e della Scienza di Torino, Torino
  - Azienda Ospedaliero-Universitaria Santa Maria della Misericordia, Udine
- Instituto Nacional de Ciencias Médicas y Nutricion Dr. Salvador Zubiran, Mexico City, Mexico City, Mexico
- Oslo Universitetssykehus HF, Ullevål, Oslo, Norway
- Poland (4):
  - COPERNICUS Podmiot Leczniczy Sp. z o. o.,, Gdansk
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Uniwersytecki Szpital Kliniczny nr 1 im. Norberta Barlickiego, Lodz
  - Samodzielny Publiczny Szpital Kliniczny Nr 4 w Lublinie, Lublin
- Serbia (3):
  - Clinical Center of Serbia, Belgrade
  - Military Medical Academy, Belgrade
  - Clinical Center Nis, Niš
- Slovakia (2):
  - Univerzitna nemocnica Bratislava Nemocnica ak. L. Derera, II. Neurologicka klinika, Bratislava
  - Fakultna nemocnica Nitra, Nitra
- Spain (4):
  - Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Universitario Virgen del Rocio, Seville
- Hallands sjukhus, Halmstad, Sweden
- Turkey (Türkiye) (5):
  - Pamukkale Uni. Med. Fac., Denizli
  - Istanbul University Cerrahpasa - Cerrahpasa Medical Faculty, Istanbul
  - Dokuz Eylul University Faculty of Medicine, Izmir
  - Selcuk Universitesi Selcuklu Tip Fakultesi Hastanesi, Konya
  - Celal Bayar University Medical Faculty, Manisa
- United Kingdom (3):
  - Southmead Hospital, Bristol, Avon
  - King's College Hospital, London, Greater London
  - The Walton Centre, Liverpool, Merseyside

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/5f6b5fc54db2bf003ab45bd5

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 54 investigative sites from December 15, 2015 to February 23, 2022. Participants with a diagnosis of Chronic Inflammatory Demyelinating Polyradiculoneuropathy (CIDP) were enrolled in this study.
Pre-assignment Details: Participants received one of the two treatments either HYQVIA/HyQvia or the 0.25% albumin placebo solution with rHuPH20 (Recombinant Human Hyaluronidase) for 6 months or until relapse in Epoch 1. Participants who relapsed during Epoch 1 received GGL/KIOVIG (participants at non-US sites) or GAMUNEX-C (participants at US sites only) in Epoch 2. A total of 138 participants were enrolled out of which 132 participants received atleast one dose of study drug.
Groups:
- Epoch 1: Placebo With rHuPH20: Participants received rHuPH20 80 U/10 mL solution, followed by SC placebo infusion at matching infusion volume as per the participant's pre-randomization monthly equivalent IG dose when administered every 2, 3, or 4 weeks for 31.54 weeks or until relapse.
- Epoch 1: HYQVIA/HyQvia: Participants received HYQVIA/HyQvia (rHuPH20) 80 U/g IG, followed by SC injection of immunoglobulin (IGI) 10% at the same monthly equivalent IG dose as per the individual participant's pre-randomized IG dose when administered every 2, 3, or 4 weeks for 30.28 weeks or until relapse.
- Epoch 2: E1: Placebo Relapse - E2: GGL/KIOVIG: Participants who were enrolled to receive placebo with rHuPH20 and achieved chronic inflammatory demyelinating polyradiculoneuropathy (CIDP) relapse during Epoch 1 received the induction dose of GGL/KIOVIG 2 g/kg bi-weekly (BW), followed by IV infusion at the same monthly equivalent dose as per the participant's pre-randomization IGIV dosing regimen when administered every 3 weeks for 25.63 weeks or until relapse.
- Epoch 2: E1: HYQVIA Relapse - E2: GGL/KIOVIG: Participants who were enrolled to receive HYQVIA/HyQvia (rHuPH20) and achieved CIDP relapse during Epoch 1 received the induction dose of GGL/KIOVIG 2 g/kg BW, followed by IV infusion at the same monthly equivalent dose as per the participant's pre-randomization IGIV dosing regimen when administered every 3 weeks for 28.67 weeks or until relapse.
- Epoch 2: E1: Placebo Relapse - E2: GAMMUNEX-C: Participants who were enrolled to receive placebo with rHuPH20 and achieved CIDP relapse during Epoch 1 received the induction dose of GAMMUNEX-C 2 g/kg BW, followed by IV infusion at the same monthly equivalent dose as per the participant's pre-randomization IGIV dosing regimen when administered every 3 weeks for 24.33 weeks or until relapse.
Period: Epoch 1: Day 1 to Approximately 32 Weeks
Arm/Group | Epoch 1: Placebo With rHuPH20 | Epoch 1: HYQVIA/HyQvia | Epoch 2: E1: Placebo Relapse - E2: GGL/KIOVIG | Epoch 2: E1: HYQVIA Relapse - E2: GGL/KIOVIG | Epoch 2: E1: Placebo Relapse - E2: GAMMUNEX-C
Started | 70 | 62 | 0 | 0 | 0
Completed | 46 | 48 | 0 | 0 | 0
Not Completed | 24 | 14 | 0 | 0 | 0
Not completed — Relapsed and Entered Epoch 2 (E2) | 17 | 4 | 0 | 0 | 0
Not completed — Relapsed and did not Enter E2 | 5 | 2 | 0 | 0 | 0
Not completed — Did not Relapse;Ended Treatment (ET) From Epoch1 | 2 | 8 | 0 | 0 | 0
Period: Epoch 2: Up to Approximately Week 61
Arm/Group | Epoch 1: Placebo With rHuPH20 | Epoch 1: HYQVIA/HyQvia | Epoch 2: E1: Placebo Relapse - E2: GGL/KIOVIG | Epoch 2: E1: HYQVIA Relapse - E2: GGL/KIOVIG | Epoch 2: E1: Placebo Relapse - E2: GAMMUNEX-C
Started | 0 | 0 | 16 | 4 | 1
Completed | 0 | 0 | 16 | 4 | 1
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Epoch 1 safety analysis set included all participants who received any study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Epoch 1: Placebo With rHuPH20 | Epoch 1: HYQVIA/HyQvia | Total
Number analyzed (Participants) | 70 | 62 | 132
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.9 (13.42) | 55.0 (14.26) | 54.4 (13.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 26 | 58
  Male | 38 | 36 | 74
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14 | 9 | 23
  Not Hispanic or Latino | 46 | 47 | 93
  Unknown or Not Reported | 10 | 6 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 3
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 64 | 58 | 122
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 3 | 7

OUTCOME MEASURES:

1. Primary Outcome: Epoch 1: Relapse Rate
Description: Relapse rate is defined as the percentage of participants who experience a worsening of functional disability. Worsening of functional disability defined as an increase of >=1 point relative to the pre- subcutaneous (SC) treatment baseline score in 2 consecutive adjusted Inflammatory Neuropathy Cause and Treatment (INCAT) disability score. The INCAT disability score is an effective and responsive tool to assess clinical response to treatment in CIDP. The disability score ranges from 0 to 10 points, where 0 is normal (eg, no upper limb problems and walking not affected) and 10 is severely incapacitated (eg, inability to move either arm for any purposeful movement and restricted to wheelchair, unable to stand and walk a few steps with help).
Time Frame: Week 32 End of Epoch 1 Treatment (EOET1)/Unscheduled relapse visit assessment (UV)/Early Termination (ET)
Population: MITT analysis set included all randomized participants who received any double-blind study medication.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Epoch 1: Placebo With rHuPH20 | Epoch 1: HYQVIA/HyQvia
Number analyzed (Participants) | 70 | 62
percentage of participants | 31.4 [21.76 to 43.03] | 9.7 [4.51 to 19.55]
Statistical Analysis 1: Comparison: Epoch 1: Placebo With rHuPH20 vs Epoch 1: HYQVIA/HyQvia; Test type: Superiority; p = 0.0045, Chi-squared; Newcombe confidence interval = -21.8, 95% CI 2-sided [-34.45 to -7.94]

2. Primary Outcome: Epoch 2: Responder Rate
Description: Responder rate is defined as clinically meaningful improvement in functional ability defined as a decrease of >=1 point in the adjusted INCAT disability score at the completion of the intravenous (IV) treatment period [6 months] or at the last study visit of the IV treatment period, relative to the pre-IV treatment baseline score.
Time Frame: Up to 6 Months post-Epoch 1 (End of Epoch 2 Treatment [EOE2T])/Unscheduled visit assessment (UV)/Early Termination
Population: E1:Placebo Relapse / E2:GGL/KIOVIG Set included a subset of participants who had a relapse while on placebo in Epoch 1, entered Epoch 2, and were treated with GAMMAGARD LIQUID/KIOVIG in Epoch 2.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Epoch 2: E1: Placebo Relapse - E2: GGL/KIOVIG: Participants who were enrolled to receive placebo with rHuPH20 and achieved CIDP relapse during Epoch 1 received the induction dose of GGL/KIOVIG 2 g/kg BW, followed by IV infusion at the same monthly equivalent dose as per the participant's pre-randomization IGIV dosing regimen when administered every 3 weeks for 25.63 weeks or until relapse.
Arm/Group | Epoch 2: E1: Placebo Relapse - E2: GGL/KIOVIG
Number analyzed (Participants) | 16
percentage of participants | 100 [80.64 to 100.00]

3. Secondary Outcome: Epoch 1: Percentage of Participants Who Experience a Worsening of Functional Disability
Description: Defined as one or more of the following: an increase of >=1 point relative to the pre-subcutaneous (SC) treatment baseline score in 2 consecutive adjusted Inflammatory Neuropathy Cause and Treatment disability scale (INCAT) scores; who experience CIDP worsening (defined as a >=8 kilo Pascal (kPa) decrease in the hand grip strength in the more affected hand); >=4 points decrease in raw Rasch-built Overall Disability Scale (R-ODS) relative to the pre-SC treatment baseline score (at the time of withdrawal from the SC treatment period). Participants are rounded off to nearest single decimal point.
Time Frame: Week 32 (EOET1)/UV/ET
Population: MITT analysis set included all randomized participants who received any double-blind study medication. Overall number of participants analyzed is the number of participants available with data.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Epoch 1: Placebo With rHuPH20 | Epoch 1: HYQVIA/HyQvia
Number analyzed (Participants) | 68 | 56
percentage of participants | 54.4 [42.66 to 65.70] | 37.5 [26.01 to 50.59]
Statistical Analysis 1: Comparison: Epoch 1: Placebo With rHuPH20 vs Epoch 1: HYQVIA/HyQvia; Test type: Superiority; p = 0.0896, Chi-squared, Corrected — The treatment groups were compared using a continuity-corrected chi-square test; Newcombe confidence interval = -16.9, 95% CI 2-sided [-33.02 to 0.69]

4. Secondary Outcome: Time to Relapse
Description: Time to relapse is defined as time from the date of the first SC administration of HYQVIA/HyQvia or placebo with rHuPH20 to the date of relapse. Participants who did not relapse were censored at their end of study.
Time Frame: Week 32 (EOET1)/UV/ET
Population: MITT analysis set included all randomized participants who received any double-blind study medication.
Measure: Median (Full Range); unit: days
Arm/Group | Epoch 1: Placebo With rHuPH20 | Epoch 1: HYQVIA/HyQvia
Number analyzed (Participants) | 70 | 62
days | NA [20 to 221] — Data for median was not estimable as less than 50% of the participants had event. | NA [7 to 217] — Data for median was not estimable as less than 50% of the participants had event.
Statistical Analysis 1: Comparison: Epoch 1: Placebo With rHuPH20 vs Epoch 1: HYQVIA/HyQvia; Test type: Superiority; p = 0.002, Wilcoxon Survival Test

5. Secondary Outcome: Epoch 1: Change From Pre-Subcutaneous (SC) Treatment Baseline in Rasch-built Overall Disability Scale (R-ODS)
Description: The Rasch-Built Overall Disability Scale (R-ODS) is a participant self-reported, linearly-weighted overall disability scale that was specifically designed to capture activity and social participation limitations in participant with immune-mediated peripheral neuropathies including CIDP. The R-ODS is comprised of 24 items for which participants are asked to rate their functioning (i.e, no difficulty, some difficulty, or could not do) related to a variety of everyday tasks at the moment of completion. The centile metric R-ODS score range is 0 to 100. Higher scores indicate better condition. The centile metric R-ODS score was used in the ANCOVA analysis. ANCOVA was used for the analysis.
Time Frame: Pre-subcutaneous (SC) treatment baseline, end of Epoch 1 treatment (approximately 7.3 months)
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Epoch 1: Placebo With rHuPH20 | Epoch 1: HYQVIA/HyQvia
Number analyzed (Participants) | 63 | 59
score on a scale | -6.1 (1.64) | -0.9 (1.69)
Statistical Analysis 1: Comparison: Epoch 1: Placebo With rHuPH20 vs Epoch 1: HYQVIA/HyQvia; Test type: Superiority; p = 0.030, ANCOVA; Least Square Mean = 5.2, 95% CI 2-sided [0.5 to 9.9]

6. Secondary Outcome: Epoch 1: Number of Participants Experiencing Any Treatment-Emergent Serious and/or Non-serious Adverse Events (SAEs and/or AEs), Regardless of Causality
Description: An AE is defined as any untoward medical occurrence in participant administered an Investigational Product (IP) that does not necessarily have a causal relationship with the treatment. An AE can therefore be any unfavorable and unintended sign (eg, an abnormal laboratory finding), symptom (eg, rash, pain, discomfort, fever, dizziness, etc.), disease (eg, peritonitis, bacteremia, etc.), or outcome of death temporally associated with the use of an IP, whether or not considered causally related to the IP. A SAE is defined as an untoward medical occurrence that at any dose meets one or more of the following criteria: outcome is fatal/results in death, is life-threatening, requires inpatient hospitalization or results in prolongation of an existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, is a medically important event, thromboembolic events, hemolytic anemia. A nonserious AE is an AE that does not meet the criteria.
Time Frame: Week 32 (EOET1)/UV/ET
Population: Epoch 1 safety analysis set included all participants who received any study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Epoch 1: Placebo With rHuPH20 | Epoch 1: HYQVIA/HyQvia
Number analyzed (Participants) | 70 | 62
Participants
  Any TEAE | 40 | 49
  Any Serious TEAE | 5 | 2

7. Secondary Outcome: Epoch 1: Number of Participants Experiencing Causally Related Serious and/or Non-Serious Adverse Events (SAEs and/or AEs)
Description: AE=any untoward medical occurrence in participant administered IP. AE can therefore be any unfavorable and unintended sign (e.g.,abnormal laboratory finding), symptom (e.g.,rash, pain, discomfort, fever, dizziness, etc.), disease (e.g.,peritonitis,bacteremia,etc.), outcome of death temporally associated with use of IP,considered causally related to the IP. SAE=untoward medical occurrence that at any dose meets following criteria: outcome is fatal/results in death, is life-threatening, requires inpatient hospitalization/results in prolongation of an existing hospitalization, results in persistent or significant disability/incapacity, is congenital anomaly/birth defect, is medically important event, thromboembolic events, hemolytic anemia. Non-SAE=AE not meeting this criteria. AE recorded by investigator as possibly/probably related to IP is considered related AE, any AE recorded as unlikely/not related is considered unrelated AE.
Time Frame: Week 32 (EOET1)/UV/ET
Population: Epoch 1 safety analysis set included all participants who received any study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Epoch 1: Placebo With rHuPH20 | Epoch 1: HYQVIA/HyQvia
Number analyzed (Participants) | 70 | 62
Participants
  Any IP-related TEAE | 19 | 38
  Any Serious IP-related TEAE | 5 | 1

8. Secondary Outcome: Epoch 1: Number of Participants With Serious and/or Non-serious Adverse Reactions (ARs) Plus Suspected ARs
Description: An AR plus suspected AR is any AE that meets any of the following criteria: an AE considered by either the investigator and/or the sponsor to be possibly or probably related to IP administration, or that begins during infusion of IP or within 72 h following the end of IP infusion, or AE for which causality assessment is missing or indeterminate. A SAE is defined as an untoward medical occurrence that at any dose meets one or more of the following criteria: outcome is fatal/results in death, is life-threatening, requires inpatient hospitalization or results in prolongation of an existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, is a medically important event, thromboembolic events, hemolytic anemia. A nonserious AE is an AE that does not meet the criteria.
Time Frame: Week 32 (EOET1)/UV/ET
Population: Epoch 1 safety analysis set included all participants who received any study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Epoch 1: Placebo With rHuPH20 | Epoch 1: HYQVIA/HyQvia
Number analyzed (Participants) | 70 | 62
Participants
  All AR/SAR | 27 | 41
  Serious AR/SAR | 5 | 1

9. Secondary Outcome: Epoch 1: Number of Treatment-emergent Serious and/or Non-serious Adverse Events (SAEs and/or AEs) Associated With Infusions Regardless of Causality
Description: AE: any untoward medical occurrence in participant administered an IP that does not necessarily have a causal relationship with the treatment. AE can therefore be any unfavorable and unintended sign (eg, an abnormal laboratory finding), symptom (eg, rash, pain, discomfort, fever, dizziness, etc.), disease (eg, peritonitis, bacteremia, etc.), or outcome of death temporally associated with the use of an IP, whether or not considered causally related to the IP. SAE: an untoward medical occurrence that at any dose meets one or more of the following criteria: outcome is fatal/results in death, is life-threatening, requires inpatient hospitalization or results in prolongation of an existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, is a medically important event, thromboembolic events, hemolytic anemia. A nonserious AE is an AE that does not meet the criteria. Participants can have more than one adverse event.
Time Frame: Week 32 (EOET1)/UV/ET
Population: Epoch 1 safety analysis set included all participants who received any study treatment. Participants can have more than one adverse event.
Measure: Number; unit: events in participants
Arm/Group | Epoch 1: Placebo With rHuPH20 | Epoch 1: HYQVIA/HyQvia
Number analyzed (Participants) | 70 | 62
events in participants
  Non-serious AEs | 144 | 340
  Serious AEs | 5 | 2

10. Secondary Outcome: Epoch 1: Number of Causally Related Serious and/or Non-serious Adverse Events (SAEs and/or AEs) Associated With Infusions
Description: AE: any untoward medical occurrence in participant administered IP. AE can therefore be any unfavorable and unintended sign (e.g., abnormal laboratory finding), symptom (e.g., rash, pain, discomfort, fever, dizziness, etc.), disease (e.g., peritonitis, bacteremia, etc.), outcome of death temporally associated with use of IP, whether or not considered causally related to the IP. SAE: untoward medical occurrence that at any dose meets following criteria: outcome is fatal/results in death, is life-threatening, requires inpatient hospitalization/results in prolongation of an existing hospitalization, results in persistent or significant disability/incapacity, is congenital anomaly/birth defect, is medically important event, (e.g., thromboembolic events, hemolytic anemia). Non-SAE:AE not meeting this criteria. AE recorded by investigator as possibly/probably related to IP is considered related AE, any AE recorded as unlikely/not related is considered unrelated AE.
Time Frame: Week 32 (EOET1)/UV/ET
Population: Epoch 1 safety analysis set included all participants who received any study treatment. Participants can have more than one causally related adverse event.
Measure: Number; unit: causally related events in participants
Arm/Group | Epoch 1: Placebo With rHuPH20 | Epoch 1: HYQVIA/HyQvia
Number analyzed (Participants) | 70 | 62
causally related events in participants
  Casually Related Non-serious Adverse Events | 53 | 223
  Casually Related Serious Adverse Events | 5 | 1

11. Secondary Outcome: Epoch 1: Number of Adverse Events (AEs) Temporally Associated With Infusions
Description: AEs occurring during an infusion or within 72 hours after completion of an infusion. An AE is defined as any untoward medical occurrence in participant administered an Investigational Product (IP) that does not necessarily have a causal relationship with the treatment. An AE can therefore be any unfavorable and unintended sign (eg, an abnormal laboratory finding), symptom (eg, rash, pain, discomfort, fever, dizziness, etc.), disease (eg, peritonitis, bacteremia, etc.), or outcome of death temporally associated with the use of an IP, whether or not considered causally related to the IP. Participants can have more than one temporally associated with infusion adverse event.
Time Frame: During an infusion or within 72 hours after completion of an infusion (up to Week 32)
Population: Epoch 1 safety analysis set included all participants who received any study treatment. Participants can have more than one temporally associated with infusion adverse event.
Measure: Number; unit: events in participants
Arm/Group | Epoch 1: Placebo With rHuPH20 | Epoch 1: HYQVIA/HyQvia
Number analyzed (Participants) | 70 | 62
events in participants | 61 | 251

12. Secondary Outcome: Epoch 1: Number of Serious and/or Non-serious Adverse Reactions (ARs) Plus Suspected ARs Associated With Infusions
Description: AR plus suspected AR: any AE that meets any of the criteria: AE considered by either investigator and/or the sponsor to be possibly or probably related to IP administration, or that begins during infusion of IP or within 72 h following end of IP infusion, or AE for which causality assessment is missing or indeterminate. SAE: untoward medical occurrence that at any dose meets one or more of following criteria: outcome is fatal/results in death, is life-threatening, requires inpatient hospitalization or results in prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, is a medically important event, thromboembolic events, hemolytic anemia. Nonserious AE is AE that does not meet the criteria. Infusion per event = number of events / total number of infusions administered (started) to participants in analysis set. Participants can have more than one AR/suspected AR associated with infusion.
Time Frame: Week 32 (EOET1)/UV/ET
Population: Epoch 1 safety analysis set included all participants who received any study treatment. Participants can have more than one AR/suspected AR associated with infusion.
Measure: Number; unit: events in participants
Arm/Group | Epoch 1: Placebo With rHuPH20 | Epoch 1: HYQVIA/HyQvia
Number analyzed (Participants) | 70 | 62
events in participants
  Non-Serious AR/Suspected AR | 76 | 261
  Serious AR/Suspected AR | 5 | 1

13. Secondary Outcome: Epoch 1: Number of Treatment-emergent Systemic Adverse Events (AEs) Associated With Infusions
Description: A treatment-emergent adverse event (TEAE) is defined as any event not present prior to the initiation of the treatments or any event already present that worsens in either intensity or frequency following exposure to the treatments. Participants can have more than one TEAE associated with infusion.
Time Frame: Week 32 (EOET1)/UV/ET
Population: Epoch 1 safety analysis set included all participants who received any study treatment. Participants can have more than one TEAE associated with infusion.
Measure: Number; unit: events in participants
Arm/Group | Epoch 1: Placebo With rHuPH20 | Epoch 1: HYQVIA/HyQvia
Number analyzed (Participants) | 70 | 62
events in participants | 149 | 342

14. Secondary Outcome: Epoch 1: Number of Treatment-emergent Local Infusion Site Reactions Associated With Infusions
Description: AE=any untoward medical occurrence in participant administered an IP that does not have causal relationship with treatment. AE can be any unfavorable and unintended sign (e.g., abnormal laboratory finding), symptom (e.g., rash, pain, discomfort, fever, dizziness, etc.), disease (e.g., peritonitis, bacteremia, etc.), or outcome of death temporally associated with the use of an IP, whether or not considered causally related to the IP. Adverse reaction/suspected adverse reaction=AE that is considered by the investigator to be possibly or probably related to IP administration, or for which the causality is indeterminate or missing, or that begins during infusion of IP or within 72 hours following the end of IP infusion. Treatment-emergent adverse events (TEAEs) are defined as adverse events that occurred during or after administration of the first dose of IP. Infusion site adverse events and injection site adverse events refer to the same type of adverse events.
Time Frame: Week 32 (EOET1)/UV/ET
Population: Epoch 1 safety analysis set included all participants who received any study treatment.
Measure: Number; unit: events in participants
Arm/Group | Epoch 1: Placebo With rHuPH20 | Epoch 1: HYQVIA/HyQvia
Number analyzed (Participants) | 70 | 62
events in participants | 20 | 141

15. Secondary Outcome: Epoch 1: Number of Infusions in Participants for Which the Infusion Rate Was Reduced And/Or the Infusion Was Interrupted or Stopped Due to Intolerability And/Or Adverse Events (AEs)
Time Frame: Week 32 (EOET1)/UV/ET
Population: Epoch 1 safety analysis set included all participants who received any study treatment.
Measure: Number; unit: number of infusions
Units Other Than Participants: number of infusions
Arm/Group | Epoch 1: Placebo With rHuPH20 | Epoch 1: HYQVIA/HyQvia
Number analyzed (Participants) | 70 | 62
Number analyzed (number of infusions) | 647 | 600
number of infusions | 1 | 3

16. Secondary Outcome: Epoch 1: Rates of Systemic and Local Adverse Events (AEs), Regardless of Causality, Expressed as Number of Events Per Infusion
Description: An AE is defined as any untoward medical occurrence in participant administered an IP that does not necessarily have a causal relationship with the treatment. An AE can therefore be any unfavorable and unintended sign (eg, an abnormal laboratory finding), symptom (eg, rash, pain, discomfort, fever, dizziness, etc.), disease (eg, peritonitis, bacteremia, etc.), or outcome of death temporally associated with the use of an IP, whether or not considered causally related to the IP. Data for number of events per infusion is assessed at the group level as follows: Per infusion = number of events / total number of infusions administered (started) to participants in the analysis set.
Time Frame: Week 32 (EOET1)/UV/ET
Population: Epoch 1 safety analysis set included all participants who received any study treatment.
Measure: Number; unit: number of AEs/infusion
Units Other Than Participants: Infusions
Arm/Group | Epoch 1: Placebo With rHuPH20 | Epoch 1: HYQVIA/HyQvia
Number analyzed (Participants) | 70 | 62
Number analyzed (Infusions) | 646 | 600
number of AEs/infusion
  Systemic Adverse Events | 0.20 | 0.34
  Local Adverse Events | 0.03 | 0.24

17. Secondary Outcome: Epoch 1: Rates of Systemic and Local Adverse Events (AEs), Regardless of Causality, Expressed as Number of Events Per Participant
Description: An AE is defined as any untoward medical occurrence in participant administered an IP that does not necessarily have a causal relationship with the treatment. An AE can therefore be any unfavorable and unintended sign (eg, an abnormal laboratory finding), symptom (eg, rash, pain, discomfort, fever, dizziness, etc.), disease (eg, peritonitis, bacteremia, etc.), or outcome of death temporally associated with the use of an IP, whether or not considered causally related to the IP. Data is reported for number of events per participant which is assessed at the group level as follows: AE per participant = number of AEs/ total number of participants in the safety analysis set.
Time Frame: Week 32 (EOET1)/UV/ET
Population: Epoch 1 safety analysis set included all participants who received any study treatment.
Measure: Number; unit: number of AEs/participant
Arm/Group | Epoch 1: Placebo With rHuPH20 | Epoch 1: HYQVIA/HyQvia
Number analyzed (Participants) | 70 | 62
number of AEs/participant
  Systemic AEs | 1.84 | 3.24
  Local AEs | 0.29 | 2.27

18. Secondary Outcome: Epoch 1: Rates of Systemic and Local Adverse Events (AEs), Regardless of Causality, Expressed as Number of Events Per 1000 Participant-year
Description: An AE is defined as any untoward medical occurrence in participant administered an IP that does not necessarily have a causal relationship with the treatment. An AE can therefore be any unfavorable and unintended sign (eg, an abnormal laboratory finding), symptom (eg, rash, pain, discomfort, fever, dizziness, etc.), disease (eg, peritonitis, bacteremia, etc.), or outcome of death temporally associated with the use of an IP, whether or not considered causally related to the IP. Data for number of events per 1000 participant-years is assessed as follows: Per 1000 participant-years = 1000 x (number of events / total number of days of exposure, i.e., the sum of duration of treatment for all participants in the safety analysis set, divided by 365.25)
Time Frame: Week 32 (EOET1)/UV/ET
Population: Epoch 1 safety analysis set included all participants who received any study treatment.
Measure: Number; unit: number of AEs/1000 participant-year
Arm/Group | Epoch 1: Placebo With rHuPH20 | Epoch 1: HYQVIA/HyQvia
Number analyzed (Participants) | 70 | 62
number of AEs/1000 participant-year
  Systemic AEs | 4689.22 | 7341.52
  Local AEs | 727.01 | 5150.02

19. Secondary Outcome: Epoch 1: Rates of Causally Related Systemic and Local Adverse Events (AEs), Expressed As Number of Events Per Infusion
Description: An AE is defined as any untoward medical occurrence in participant administered an IP that does not necessarily have a causal relationship with the treatment. An AE can therefore be any unfavorable and unintended sign (eg, an abnormal laboratory finding), symptom (eg, rash, pain, discomfort, fever, dizziness, etc.), disease (eg, peritonitis, bacteremia, etc.), or outcome of death temporally associated with the use of an IP, whether or not considered causally related to the IP. An AE that is recorded by the investigator as possibly related or probably related to IP was considered a related AE, and any AE recorded as unlikely related or not related was considered unrelated AE. Data for number of events per infusion is assessed at the group level as follows: Per infusion = number of events / total number of infusions administered (started) to participants in the analysis set.
Time Frame: Week 32 (EOET1)/UV/ET
Population: Epoch 1 safety analysis set included all participants who received any study treatment.
Measure: Number; unit: number of AEs/infusion
Units Other Than Participants: Infusions
Arm/Group | Epoch 1: Placebo With rHuPH20 | Epoch 1: HYQVIA/HyQvia
Number analyzed (Participants) | 70 | 62
Number analyzed (Infusions) | 646 | 600
number of AEs/infusion
  IP-Related Systemic TEAE | 0.06 | 0.17
  IP-Related Local TEAE | 0.02 | 0.21

20. Secondary Outcome: Epoch 1: Rates of Causally Related Systemic and Local Adverse Events (AEs), Expressed As Number of Events Per Participant
Description: An AE is defined as any untoward medical occurrence in participant administered an IP that does not necessarily have a causal relationship with the treatment. An AE can therefore be any unfavorable and unintended sign (eg, an abnormal laboratory finding), symptom (eg, rash, pain, discomfort, fever, dizziness, etc.), disease (eg, peritonitis, bacteremia, etc.), or outcome of death temporally associated with the use of an IP, whether or not considered causally related to the IP. An AE that is recorded by the investigator as possibly related or probably related to IP was considered a related AE, and any AE recorded as unlikely related or not related was considered unrelated AE. Data is reported for number of events per participant which is assessed at the group level as follows: AE per participant = number of AEs/ total number of participants in the safety analysis set.
Time Frame: Week 32 (EOET1)/UV/ET
Population: Epoch 1 safety analysis set included all participants who received any study treatment.
Measure: Number; unit: number of AEs/participant
Arm/Group | Epoch 1: Placebo With rHuPH20 | Epoch 1: HYQVIA/HyQvia
Number analyzed (Participants) | 70 | 62
number of AEs/participant
  IP-related Systemic TEAE | 0.54 | 1.6
  IP-related Local TEAE | 0.21 | 2

21. Secondary Outcome: Epoch 1: Rates of Causally Related Systemic and Local Adverse Events (AEs), Expressed as Number of Events Per Participant-year
Description: An AE is defined as any untoward medical occurrence in participant administered an IP that does not necessarily have a causal relationship with the treatment. An AE can therefore be any unfavorable and unintended sign (eg, an abnormal laboratory finding), symptom (eg, rash, pain, discomfort, fever, dizziness, etc.), disease (eg, peritonitis, bacteremia, etc.), or outcome of death temporally associated with the use of an IP, whether or not considered causally related to the IP. An AE that is recorded by the investigator as possibly related or probably related to IP was considered a related AE, and any AE recorded as unlikely related or not related was considered unrelated AE.
Time Frame: Week 32 (EOET1)/UV/ET
Population: Epoch 1 safety analysis set included all participants who received any study treatment.
Measure: Number; unit: number of AEs/1000 participant-year
Arm/Group | Epoch 1: Placebo With rHuPH20 | Epoch 1: HYQVIA/HyQvia
Number analyzed (Participants) | 70 | 62
number of AEs/1000 participant-year
  IP-related Systemic TEAE | 1381.32 | 3615.98
  IP-related Local TEAE | 545.26 | 4529.1

22. Secondary Outcome: Epoch 1: Rates of Systemic and Local Adverse Reactions (ARs) Plus Suspected ARs, Expressed as Number of Events Per Infusion
Description: An AR plus suspected AR is any AE that meets any of the following criteria: an AE considered by either the investigator and/or the sponsor to be possibly or probably related to IP administration, or that begins during infusion of IP or within 72 h following the end of IP infusion, or AE for which causality assessment is missing or indeterminate. Data for number of events per infusion is assessed at the group level as follows: Per infusion = number of events / total number of infusions administered (started) to participants in the analysis set.
Time Frame: Week 32 (EOET1)/UV/ET
Population: Epoch 1 safety analysis set included all participants who received any study treatment.
Measure: Number; unit: number of ARs/infusion
Units Other Than Participants: Infusions
Arm/Group | Epoch 1: Placebo With rHuPH20 | Epoch 1: HYQVIA/HyQvia
Number analyzed (Participants) | 70 | 62
Number analyzed (Infusions) | 646 | 600
number of ARs/infusion
  Systemic Plus Suspected ARs | 0.09 | 0.20
  Local Plus Suspected ARs | 0.03 | 0.24

23. Secondary Outcome: Epoch 1: Rates of Systemic and Local Adverse Reactions (ARs) Plus Suspected ARs, Expressed as Number of Events Per Participant
Description: An AR plus suspected AR is any AE that meets any of the following criteria: an AE considered by either the investigator and/or the sponsor to be possibly or probably related to IP administration, or that begins during infusion of IP or within 72 h following the end of IP infusion, or AE for which causality assessment is missing or indeterminate. Data is reported for number of events per participant which is assessed at the group level as follows: AE per participant = number of AEs/ total number of participants in the safety analysis set.
Time Frame: Week 32 (EOET1)/UV/ET
Population: Epoch 1 safety analysis set included all participants who received any study treatment.
Measure: Number; unit: number of ARs/participant
Arm/Group | Epoch 1: Placebo With rHuPH20 | Epoch 1: HYQVIA/HyQvia
Number analyzed (Participants) | 70 | 62
number of ARs/participant
  Systemic Plus Suspected ARs | 0.80 | 1.94
  Local Plus Suspected ARs | 0.29 | 2.27

24. Secondary Outcome: Epoch 1: Rates of Systemic and Local Adverse Reactions (ARs) Plus Suspected ARs, Expressed as Number of Events Per 1000 Participant-Year
Description: An AR plus suspected AR is any AE that meets any of the following criteria: an AE considered by either the investigator and/or the sponsor to be possibly or probably related to IP administration, or that begins during infusion of IP or within 72 h following the end of IP infusion, or AE for which causality assessment is missing or indeterminate. Data for number of events per 1000 participant-years is assessed as follows: Per 1000 participant-years = 1000 x (number of events / total number of days of exposure, i.e., the sum of duration of treatment for all participants in the safety analysis set, divided by 365.25)
Time Frame: Week 32 (EOET1)/UV/ET
Population: Epoch 1 safety analysis set included all participants who received any study treatment.
Measure: Number; unit: number of ARs/1000 Participant year
Arm/Group | Epoch 1: Placebo With rHuPH20 | Epoch 1: HYQVIA/HyQvia
Number analyzed (Participants) | 70 | 62
number of ARs/1000 Participant year
  Systemic Plus Suspected ARs | 2035.63 | 4383.00
  Local Plus Suspected ARs | 727.01 | 5150.02

25. Secondary Outcome: Epoch 1: Number of Participants Who Develop Binding and/or Neutralizing Antibodies to Recombinant Human Hyaluronidase (rHuPH20)
Description: Number of participants who developed binding and/or neutralizing antibodies to rHuPH20 in Epoch 1 were reported. High-binding antibodies is defined as number of participants who had at least one anti-rHuPH20 antibody titer ≥1:160 during treatment.
Time Frame: Week 32 (EOET1)/UV/ET
Population: Epoch 1 safety analysis set included all participants who received any study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Epoch 1: Placebo With rHuPH20 | Epoch 1: HYQVIA/HyQvia
Number analyzed (Participants) | 70 | 62
Participants | 7 | 1

26. Secondary Outcome: Epoch 2: Number of Participants Experiencing Any Treatment-emergent Serious and/or Non-serious Adverse Events (SAEs and/or AEs), Regardless of Causality
Description: Number of participants experiencing any treatment-emergent serious and/or non-serious adverse events regardless of causality in Epoch 2 was reported.
Time Frame: Throughout Epoch 2, up to 6 months post-Epoch 1
Population: Epoch 2 safety analysis set included all participants who had a relapse in Epoch 1, entered Epoch 2, and received IGIV treatment with either GGL/KIOVIG or GAMUNEX-C.
Measure: Count of Participants; unit: Participants
Arm/Group | Epoch 2: E1: Placebo Relapse - E2: GGL/KIOVIG | Epoch 2: E1: HYQVIA Relapse - E2: GGL/KIOVIG | Epoch 2: E1: Placebo Relapse - E2: GAMMUNEX-C
Number analyzed (Participants) | 16 | 4 | 1
Participants
  Any IP related TEAE | 11 | 3 | 1
  Any IP related serious TEAE | 0 | 0 | 0

27. Secondary Outcome: Epoch 2: Number of Participants Experiencing Causally Related Serious and/or Non-serious Adverse Events (SAEs and/or AEs)
Description: as for outcome 10
Time Frame: Throughout Epoch 2, up to 6 months post-Epoch 1
Population: as for outcome 26
Measure: Count of Participants; unit: Participants
Arm/Group | Epoch 2: E1: Placebo Relapse - E2: GGL/KIOVIG | Epoch 2: E1: HYQVIA Relapse - E2: GGL/KIOVIG | Epoch 2: E1: Placebo Relapse - E2: GAMMUNEX-C
Number analyzed (Participants) | 16 | 4 | 1
Participants
  Causally related AEs | 8 | 3 | 0
  Causally related SAEs | 0 | 0 | 0

28. Secondary Outcome: Epoch 2: Number of Participants With Serious and/or Non-serious Adverse Reactions (ARs) Plus Suspected ARs
Description: An adverse reaction/suspected adverse reaction is defined as an Adverse Event that is considered by the investigator to be possibly or probably related to IP administration, or for which the causality is indeterminate or missing, or that begins during infusion of IP or within 72 hours following the end of IP infusion.
Time Frame: Throughout Epoch 2, up to 6 months post-Epoch 1
Population: as for outcome 26
Measure: Count of Participants; unit: Participants
Arm/Group | Epoch 2: E1: Placebo Relapse - E2: GGL/KIOVIG | Epoch 2: E1: HYQVIA Relapse - E2: GGL/KIOVIG | Epoch 2: E1: Placebo Relapse - E2: GAMMUNEX-C
Number analyzed (Participants) | 16 | 4 | 1
Participants
  Any AR/SAR | 10 | 3 | 0
  Any Serious AR/SAR | 0 | 0 | 0

29. Secondary Outcome: Epoch 2: Number of Treatment-emergent Serious and/or Non-serious Adverse Events (SAEs and/or AEs) Associated With Infusions Regardless of Causality
Description: A SAE is defined as an untoward medical occurrence that at any dose meets one or more of the following criteria: outcome is fatal/results in death, is life-threatening, requires inpatient hospitalization or results in prolongation of an existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, is a medically important event, thromboembolic events, hemolytic anemia. A nonserious AE is an AE that does not meet the criteria. An AR plus suspected AR is any AE that meets any of the following criteria: an AE considered by either the investigator and/or the sponsor to be possibly or probably related to IP administration, or that begins during infusion of IP or within 72 h following the end of IP infusion, or AE for which causality assessment is missing or indeterminate. Participants can have more than one adverse event.
Time Frame: Throughout Epoch 2, up to 6 months post-Epoch 1
Population: Epoch 2 safety analysis set included all participants who had a relapse in Epoch 1, entered Epoch 2, and received IGIV treatment with either GGL/KIOVIG or GAMUNEX-C. Participants can have more than one adverse event.
Measure: Number; unit: events in participants
Arm/Group | Epoch 2: E1: Placebo Relapse - E2: GGL/KIOVIG | Epoch 2: E1: HYQVIA Relapse - E2: GGL/KIOVIG | Epoch 2: E1: Placebo Relapse - E2: GAMMUNEX-C
Number analyzed (Participants) | 16 | 4 | 1
events in participants
  Serious AEs | 0 | 0 | 0
  Non-serious AEs | 35 | 25 | 1

30. Secondary Outcome: Epoch 2: Number of Causally Related Serious and/or Non-serious Adverse Events (SAEs and/or AEs) Associated With Infusions
Description: as for outcome 10
Time Frame: Throughout Epoch 2, up to 6 months post-Epoch 1
Population: as for outcome 29
Measure: Number; unit: events in participants
Arm/Group | Epoch 2: E1: Placebo Relapse - E2: GGL/KIOVIG | Epoch 2: E1: HYQVIA Relapse - E2: GGL/KIOVIG | Epoch 2: E1: Placebo Relapse - E2: GAMMUNEX-C
Number analyzed (Participants) | 16 | 4 | 1
events in participants
  Any TEAE | 23 | 0 | 0
  Any serious TEAE | 0 | 0 | 0

31. Secondary Outcome: Epoch 2: Number of Adverse Events (AEs) Temporally Associated With Infusions
Description: AEs occurring during an infusion or within 72 hours after completion of an infusion. An AE is defined as any untoward medical occurrence in participant administered an IP that does not necessarily have a causal relationship with the treatment. An AE can therefore be any unfavorable and unintended sign (eg, an abnormal laboratory finding), symptom (eg, rash, pain, discomfort, fever, dizziness, etc.), disease (eg, peritonitis, bacteremia, etc.), or outcome of death temporally associated with the use of an IP, whether or not considered causally related to the IP. Participants can have more than one adverse event.
Time Frame: During an infusion or within 72 hours after completion of an infusion (up to Week 32)
Population: as for outcome 29
Measure: Number; unit: events in participants
Arm/Group | Epoch 2: E1: Placebo Relapse - E2: GGL/KIOVIG | Epoch 2: E1: HYQVIA Relapse - E2: GGL/KIOVIG | Epoch 2: E1: Placebo Relapse - E2: GAMMUNEX-C
Number analyzed (Participants) | 16 | 4 | 1
events in participants | 25 | 11 | 0

32. Secondary Outcome: Epoch 2: Number of Serious and/or Non-serious Adverse Reactions (ARs) Plus Suspected ARs Associated With Infusions
Description: A SAE is defined as an untoward medical occurrence that at any dose meets one or more of the following criteria: outcome is fatal/results in death, is life-threatening, requires inpatient hospitalization or results in prolongation of an existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, is a medically important event, thromboembolic events, hemolytic anemia. A nonserious AE is an AE that does not meet the criteria. An AR plus suspected AR is any AE that meets any of the following criteria: an AE considered by either the investigator and/or the sponsor to be possibly or probably related to IP administration, or that begins during infusion of IP or within 72 h following the end of IP infusion, or AE for which causality assessment is missing or indeterminate. Participants can have more than one AR/SAR.
Time Frame: Throughout Epoch 2, up to 6 months post-Epoch 1
Population: Epoch 2 safety analysis set included all participants who had a relapse in Epoch 1, entered Epoch 2, and received IGIV treatment with either GGL/KIOVIG or GAMUNEX-C. Participants can have more than one AR/SAR.
Measure: Number; unit: events in participants
Arm/Group | Epoch 2: E1: Placebo Relapse - E2: GGL/KIOVIG | Epoch 2: E1: HYQVIA Relapse - E2: GGL/KIOVIG | Epoch 2: E1: Placebo Relapse - E2: GAMMUNEX-C
Number analyzed (Participants) | 16 | 4 | 1
events in participants
  AR/SAR | 28 | 11 | 0
  Serious AR/SAR | 0 | 0 | 0

33. Secondary Outcome: Epoch 2: Number of Treatment-emergent Systemic Adverse Events (AEs) Associated With Infusions
Description: A treatment-emergent adverse event (TEAE) is defined as any event not present prior to the initiation of the treatments or any event already present that worsens in either intensity or frequency following exposure to the treatments. Participants can have more than one treatment-emergent systemic AEs.
Time Frame: Throughout Epoch 2, up to 6 months post-Epoch 1
Population: Epoch 2 safety analysis set included all participants who had a relapse in Epoch 1, entered Epoch 2, and received IGIV treatment with either GGL/KIOVIG or GAMUNEX-C. Participants can have more than one treatment-emergent systemic AEs.
Measure: Number; unit: events in participants
Arm/Group | Epoch 2: E1: Placebo Relapse - E2: GGL/KIOVIG | Epoch 2: E1: HYQVIA Relapse - E2: GGL/KIOVIG | Epoch 2: E1: Placebo Relapse - E2: GAMMUNEX-C
Number analyzed (Participants) | 16 | 4 | 1
events in participants | 35 | 25 | 1

34. Secondary Outcome: Epoch 2: Number of Treatment-emergent Local Infusion Site Reactions Associated With Infusions
Description: AE=any untoward medical occurrence in participant administered an IP that does not have causal relationship with treatment. AE can be any unfavorable and unintended sign (e.g., abnormal laboratory finding), symptom (e.g., rash, pain, discomfort, fever, dizziness, etc.), disease (e.g., peritonitis, bacteremia, etc.), or outcome of death temporally associated with the use of an IP, whether or not considered causally related to the IP. Adverse reaction/suspected adverse reaction=AE that is considered by the investigator to be possibly or probably related to IP administration, or for which the causality is indeterminate or missing, or that begins during infusion of IP or within 72 hours following the end of IP infusion. TEAEs are defined as adverse events that occurred during or after administration of the first dose of IP. Infusion site adverse events and injection site adverse events refer to the same type of adverse events.
Time Frame: Throughout Epoch 2, up to 6 months post-Epoch 1
Population: as for outcome 26
Measure: Number; unit: events in participants
Arm/Group | Epoch 2: E1: Placebo Relapse - E2: GGL/KIOVIG | Epoch 2: E1: HYQVIA Relapse - E2: GGL/KIOVIG | Epoch 2: E1: Placebo Relapse - E2: GAMMUNEX-C
Number analyzed (Participants) | 16 | 4 | 1
events in participants | 0 | 0 | 0

35. Secondary Outcome: Epoch 2: Number of Infusions for Which the Infusion Rate Was Reduced and/or the Infusion Was Interrupted or Stopped Due to Intolerability and/or Adverse Events (AEs)
Description: An AE is defined as any untoward medical occurrence in participant administered an IP that does not necessarily have a causal relationship with the treatment. An AE can therefore be any unfavorable and unintended sign (eg, an abnormal laboratory finding), symptom (eg, rash, pain, discomfort, fever, dizziness, etc.), disease (eg, peritonitis, bacteremia, etc.), or outcome of death temporally associated with the use of an IP, whether or not considered causally related to the IP.
Time Frame: Throughout Epoch 2, up to 6 months post-Epoch 1
Population: Epoch 2 IGIV Analysis Set included participants who relapsed in Epoch 1 and received at least one dose of IGIV treatment (GGL/KIOVIG or GAMMUNEX-C).
Measure: Number; unit: number of infusions
Units Other Than Participants: number of infusions
Arm/Group | Epoch 2: E1: Placebo Relapse - E2: GGL/KIOVIG | Epoch 2: E1: HYQVIA Relapse - E2: GGL/KIOVIG
Number analyzed (Participants) | 16 | 4
Number analyzed (number of infusions) | 328 | 61
number of infusions | 1 | 1

36. Secondary Outcome: Epoch 2: Rates of Systemic and Local Adverse Events (AEs), Regardless of Causality, Expressed as Number of Events Per Infusion
Description: as for outcome 16
Time Frame: Throughout Epoch 2, up to 6 months post-Epoch 1
Population: as for outcome 26
Measure: Number; unit: number of AEs/infusion
Units Other Than Participants: Infusions
Arm/Group | Epoch 2: E1: Placebo Relapse - E2: GGL/KIOVIG | Epoch 2: E1: HYQVIA Relapse - E2: GGL/KIOVIG | Epoch 2: E1: Placebo Relapse - E2: GAMMUNEX-C
Number analyzed (Participants) | 16 | 4 | 1
Number analyzed (Infusions) | 328 | 61 | 18
number of AEs/infusion
  Systemic AEs | 0.11 | 0.41 | 0.06
  Local AEs | 0 | 0 | 0

37. Secondary Outcome: Epoch 2: Rates of Systemic and Local Adverse Events (AEs), Regardless of Causality, Expressed as Number of Events Per Participant
Description: as for outcome 17
Time Frame: Throughout Epoch 2, up to 6 months post-Epoch 1
Population: as for outcome 26
Measure: Number; unit: number of AEs/participant
Arm/Group | Epoch 2: E1: Placebo Relapse - E2: GGL/KIOVIG | Epoch 2: E1: HYQVIA Relapse - E2: GGL/KIOVIG | Epoch 2: E1: Placebo Relapse - E2: GAMMUNEX-C
Number analyzed (Participants) | 16 | 4 | 1
number of AEs/participant
  Systemic AEs | 2.19 | 6.25 | 1.00
  Local AEs | 0 | 0 | 0

38. Secondary Outcome: Epoch 2: Rates of Systemic and Local Adverse Events (AEs), Regardless of Causality, Expressed as Number of Events Per 1000 Participant-year
Description: as for outcome 35
Time Frame: Throughout Epoch 2, up to 6 months post-Epoch 1
Population: as for outcome 26
Measure: Number; unit: number of AEs/1000 participant-year
Arm/Group | Epoch 2: E1: Placebo Relapse - E2: GGL/KIOVIG | Epoch 2: E1: HYQVIA Relapse - E2: GGL/KIOVIG | Epoch 2: E1: Placebo Relapse - E2: GAMMUNEX-C
Number analyzed (Participants) | 16 | 4 | 1
number of AEs/1000 participant-year
  Systemic AEs | 4645.26 | 12806.80 | 2135.96
  Local AEs | 0 | 0 | 0

39. Secondary Outcome: Epoch 2: Rates of Causally Related Systemic and Local Adverse Events (AEs), Expressed As Number of Events Per Infusion
Description: as for outcome 19
Time Frame: Throughout Epoch 2, up to 6 months post-Epoch 1
Population: as for outcome 26
Measure: Number; unit: number of AEs/infusion
Units Other Than Participants: Infusions
Arm/Group | Epoch 2: E1: Placebo Relapse - E2: GGL/KIOVIG | Epoch 2: E1: HYQVIA Relapse - E2: GGL/KIOVIG | Epoch 2: E1: Placebo Relapse - E2: GAMMUNEX-C
Number analyzed (Participants) | 16 | 4 | 1
Number analyzed (Infusions) | 328 | 61 | 18
number of AEs/infusion
  IP-related Systemic Adverse Events | 0.07 | 0.13 | 0
  IP-related Local Adverse Events | 0 | 0 | 0

40. Secondary Outcome: Epoch 2: Rates of Causally Related Systemic and Local Adverse Events (AEs), Expressed as Number of Events Per Participant
Description: as for outcome 20
Time Frame: Throughout Epoch 2, up to 6 months post-Epoch 1
Population: as for outcome 26
Measure: Number; unit: number of AEs/participant
Arm/Group | Epoch 2: E1: Placebo Relapse - E2: GGL/KIOVIG | Epoch 2: E1: HYQVIA Relapse - E2: GGL/KIOVIG | Epoch 2: E1: Placebo Relapse - E2: GAMMUNEX-C
Number analyzed (Participants) | 16 | 4 | 1
number of AEs/participant
  IP-related Systemic Adverse Events | 1.44 | 2 | 0
  IP-related Local Adverse Events | 0 | 0 | 0

41. Secondary Outcome: Epoch 2: Rates of Causally Related Systemic and Local Adverse Events (AEs), Expressed as Number of Events Per Participant-Year
Description: as for outcome 21
Time Frame: Throughout Epoch 2, up to 6 months post-Epoch 1
Population: as for outcome 26
Measure: Number; unit: number of AEs/1000 participant-year
Arm/Group | Epoch 2: E1: Placebo Relapse - E2: GGL/KIOVIG | Epoch 2: E1: HYQVIA Relapse - E2: GGL/KIOVIG | Epoch 2: E1: Placebo Relapse - E2: GAMMUNEX-C
Number analyzed (Participants) | 16 | 4 | 1
number of AEs/1000 participant-year
  IP-related Systemic Adverse Events | 3052.6 | 4098.18 | 0
  IP-related Local Adverse Events | 0 | 0 | 0

42. Secondary Outcome: Epoch 2: Rates of Systemic and Local Adverse Reactions (ARs) Plus Suspected Ars, Expressed as Number of Events Per Infusion
Description: as for outcome 22
Time Frame: Throughout Epoch 2, up to 6 months post-Epoch 1
Population: as for outcome 26
Measure: Number; unit: number of ARs/infusion
Units Other Than Participants: Infusions
Arm/Group | Epoch 2: E1: Placebo Relapse - E2: GGL/KIOVIG | Epoch 2: E1: HYQVIA Relapse - E2: GGL/KIOVIG | Epoch 2: E1: Placebo Relapse - E2: GAMMUNEX-C
Number analyzed (Participants) | 16 | 4 | 1
Number analyzed (Infusions) | 328 | 16 | 18
number of ARs/infusion
  Systemic plus Suspected ARs | 0.09 | 0.18 | 0
  Local plus Suspected ARs | 0 | 0 | 0

43. Secondary Outcome: Epoch 2: Rates of Systemic and Local Adverse Reactions (ARs) Plus Suspected ARs, Expressed as Number of Events Per Participant
Description: as for outcome 23
Time Frame: Throughout Epoch 2, up to 6 months post-Epoch 1
Population: as for outcome 26
Measure: Number; unit: number of ARs/participant
Arm/Group | Epoch 2: E1: Placebo Relapse - E2: GGL/KIOVIG | Epoch 2: E1: HYQVIA Relapse - E2: GGL/KIOVIG | Epoch 2: E1: Placebo Relapse - E2: GAMMUNEX-C
Number analyzed (Participants) | 16 | 4 | 1
number of ARs/participant
  Systemic plus Suspected ARs | 1.75 | 2.75 | 0
  Local plus Suspected ARs | 0 | 0 | 0

44. Secondary Outcome: Epoch 2: Rates of Systemic and Local Adverse Reactions (ARs) Plus Suspected ARs, Expressed as Number of Events Per 1000 Participant-Year
Description: as for outcome 24
Time Frame: Throughout Epoch 2, up to 6 months post-Epoch 1
Population: as for outcome 26
Measure: Number; unit: number of ARs/1000 participant-year
Arm/Group | Epoch 2: E1: Placebo Relapse - E2: GGL/KIOVIG | Epoch 2: E1: HYQVIA Relapse - E2: GGL/KIOVIG | Epoch 2: E1: Placebo Relapse - E2: GAMMUNEX-C
Number analyzed (Participants) | 16 | 4 | 1
number of ARs/1000 participant-year
  Systemic plus Suspected ARs | 3716.21 | 5634.99 | 0
  Local plus Suspected ARs | 0 | 0 | 0

45. Secondary Outcome: Epoch 2: Percentage of Participants With Clinically Meaningful Improvement in Functional Ability
Description: Defined as one or more of the following: a decrease of >=1 point in the adjusted Inflammatory Neuropathy Cause and Treatment disability scale (INCAT) score at 2 consecutive time points; who experience CIDP improvement (defined as ≥8 kilo Pascal (kPa) increase in hand grip strength in the more affected hand; >=4 points increase in Rasch-built Overall Disability Scale (R-ODS)) at the completion of the intravenous (IV) treatment period [6 months] or at the last study visit of the IV treatment period, relative to the pre-IV treatment baseline score.
Time Frame: Throughout Epoch 2, up to 6 months post-Epoch 1
Population: as for outcome 35
Measure: Number; unit: percentage of participants
Groups:
- Epoch 2: E1: Placebo Relapse - E2: IGIV: Participants who were enrolled to receive placebo with rHuPH20 and achieved CIDP relapse during Epoch 1 received the induction dose of GGL/KIOVIG or GAMMUNEX-C 2 g/kg BW, followed by IV infusion at the same monthly equivalent dose as per the participant's pre-randomization IGIV dosing regimen when administered every 3 weeks for 25.63 weeks or until relapse.
- Epoch 2: E1: HYQVIA Relapse - E2: IGIV: Participants who were enrolled to receive HYQVIA/HyQvia (rHuPH20) and achieved CIDP relapse during Epoch 1 received the induction dose of GGL/KIOVIG 2 g/kg BW, followed by IV infusion at the same monthly equivalent dose as per the participant's pre-randomization IGIV dosing regimen when administered every 3 weeks for 28.67 weeks or until relapse.
Arm/Group | Epoch 2: E1: Placebo Relapse - E2: IGIV | Epoch 2: E1: HYQVIA Relapse - E2: IGIV
Number analyzed (Participants) | 17 | 4
percentage of participants | 100 [80.64 to 100] | 100 [NA to NA]

ADVERSE EVENTS:
Time Frame: From the date of signing of the informed consent form up to the end of the study, approximately 74 months.
Description: Epoch 1 safety analysis set included all participants who received any study treatment. Epoch 2 safety analysis set included all participants who had a relapse in Epoch 1, entered Epoch 2, and received IGIV treatment with either GGL/KIOVIG or GAMUNEX-C.
Arm/Group | Epoch 1: Placebo With rHuPH20 | Epoch 1: HYQVIA/HyQvia | Epoch 2: E1: Placebo Relapse - E2: GGL/KIOVIG | Epoch 2: E1: HYQVIA Relapse - E2: GGL/KIOVIG | Epoch 2: E1: Placebo Relapse - E2: GAMMUNEX-C
All-Cause Mortality (participants affected / at risk) | 0/70 | 0/62 | 0/16 | 0/4 | 0/1
Serious Adverse Events (participants affected / at risk) | 5/70 | 2/62 | 0/16 | 0/4 | 0/1
Other Adverse Events (participants affected / at risk) | 19/70 | 42/62 | 11/16 | 3/4 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Epoch 1: Placebo With rHuPH20 (N=70) | Epoch 1: HYQVIA/HyQvia (N=62) | Epoch 2: E1: Placebo Relapse - E2: GGL/KIOVIG (N=16) | Epoch 2: E1: HYQVIA Relapse - E2: GGL/KIOVIG (N=4) | Epoch 2: E1: Placebo Relapse - E2: GAMMUNEX-C (N=1)
Arrhythmia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Chronic inflammatory demyelinating polyradiculoneuropathy (Nervous system disorders) | 4 | 0 | 0 | 0 | 0
Otitis media chronic (Infections and infestations) | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Epoch 1: Placebo With rHuPH20 (N=70) | Epoch 1: HYQVIA/HyQvia (N=62) | Epoch 2: E1: Placebo Relapse - E2: GGL/KIOVIG (N=16) | Epoch 2: E1: HYQVIA Relapse - E2: GGL/KIOVIG (N=4) | Epoch 2: E1: Placebo Relapse - E2: GAMMUNEX-C (N=1)
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 4 | 0 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 1
Blood creatinine increased (Investigations) | 0 | 0 | 1 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 1 | 0 | 0
Chills (General disorders) | 0 | 1 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 5 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 4 | 1 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 2 | 6 | 1 | 0 | 0
Headache (Nervous system disorders) | 8 | 8 | 6 | 2 | 0
Hypertension (Vascular disorders) | 1 | 4 | 0 | 0 | 0
Illness (General disorders) | 0 | 0 | 1 | 0 | 0
Infusion site erythema (General disorders) | 0 | 6 | 0 | 0 | 0
Infusion site oedema (General disorders) | 1 | 4 | 0 | 0 | 0
Infusion site pain (General disorders) | 2 | 5 | 0 | 0 | 0
Infusion site pruritus (General disorders) | 0 | 4 | 0 | 0 | 0
Injection site erythema (General disorders) | 0 | 7 | 0 | 0 | 0
Injection site pain (General disorders) | 2 | 5 | 0 | 0 | 0
Injection site pruritus (General disorders) | 0 | 4 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 0 | 0
Migraine (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 1 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 7 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 3 | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 5 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 7 | 1 | 1 | 0
Somnolence (Nervous system disorders) | 0 | 1 | 1 | 0 | 0
Tremor (Nervous system disorders) | 0 | 2 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 4 | 1 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Study Protocol (2021-05-20): https://cdn.clinicaltrials.gov/large-docs/70/NCT02549170/Prot_000.pdf
  • Statistical Analysis Plan (2022-04-25): https://cdn.clinicaltrials.gov/large-docs/70/NCT02549170/SAP_001.pdf